CLINICAL TRIAL: NCT01195753
Title: Open, Prospective, Historic-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Infusion of Liver Cell Suspension (HHLivC) in Children With Urea Cycle Disorders.
Brief Title: Human Heterologous Liver Cells for Infusion in Children With Urea Cycle Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cytonet GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD05
Record Dates: First submitted 2010-03-02; First posted 2010-09-06 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Urea Cycle Disorders
Keywords: Urea cycle Disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liver Cell Infusion (Experimental)
  Interventions: Biological: HHLivC

INTERVENTIONS:
Biological: HHLivC — multiple infusion of liver cells

SUMMARY:
Treatment with liver cell infusion for children with urea cycle disorders (UCD).

DETAILED DESCRIPTION:
Urea cycle disorders are rare inherited diseases that generally have a poor outcome, especially with onset of the disease in the neonatal period. UCDs are caused by a deficiency of one of six enzymes responsible for removing ammonia from the bloodstream. Instead of being converted into urea which is removed from the body with the urine, ammonia accumulates in UCD patients leading to brain damage or death. In the light of a mortality rate of > 50% at the age of 10 years the current pharmacological and dietary therapy is of modest success. Furthermore, mental retardation, cerebral palsy and other neurological sequelae are common among surviving patients.

In the last years, orthotopic liver transplantation (OLT) has become the best therapeutic option for UCD with long-term survival rates of about 90%. However, in the first weeks of life OLT still is technically demanding and prone to complications. With larger size of the recipient, the technical problems with OLT decrease considerably. The increased body weight usually achieved at the age of more than 8 weeks is related to a major reduction in transplantation related morbidity. Stabilization of metabolism until the patient can undergo OLT is essential.

In this study, young children with UCD will be treated by repetitive application of human liver cells. In the last consequence, the aim of this new therapy option is to supply a sufficient amount of healthy liver cells to compensate for the metabolic defect and to reduce the risk of neurological deterioration while awaiting OLT.

ELIGIBILITY:
Inclusion Criteria:

* Age: birth up to 5 years of age
* Ornithine transcarbamylase deficiency [OTCD], Carbamyl phosphate synthetase I deficiency [CPSD], Argininosuccinate synthetase deficiency [ASSD, Citrullinaemia]
* Written Informed Consent

Exclusion Criteria:

* Weight ≤ 3.5 kg
* Presence of acute infection at the time of inclusion
* Severe chronic or systemic disease other than study indication
* Structural liver disease (eg, cirrhosis, portal hypertension)
* Required valproate therapy

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in 13C urea formation from baseline to 2 and 4 months after first HHLivC infusion | Baseline to 2 and 4 months

SECONDARY OUTCOMES:
Frequency and severity of metabolic crises | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Stanford University, Palo Alto, California
  - University of California, San Diego, California
  - Yale University, New Haven, Connecticut
  - Children's Memorial Hospital, Chicago, Illinois
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Meyburg J, Das AM, Hoerster F, Lindner M, Kriegbaum H, Engelmann G, Schmidt J, Ott M, Pettenazzo A, Luecke T, Bertram H, Hoffmann GF, Burlina A. One liver for four children: first clinical series of liver cell transplantation for severe neonatal urea cycle defects. Transplantation. 2009 Mar 15;87(5):636-41. doi: 10.1097/TP.0b013e318199936a. PMID 19295306